CLINICAL TRIAL: NCT03376737
Title: A Single-Arm Phase II Clinical Trial of Apatinib as the Maintenance Therapy in Advanced Lung Adenocarcinoma
Brief Title: Study of Apatinib as the Maintenance Therapy in Advanced Lung Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HNP012
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — apatinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib + Pemetrexed (Experimental): Apatinib + Pemetrexed
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib (250 mg/d) + Pemetrexed (500 mg/m2)
  Other Names: Pemetrexed

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Apatinib plus Pemetrexed as the Maintenance Therapy in Advanced Lung Adenocarcinoma.

DETAILED DESCRIPTION:
Lung adenocarcinoma is the most common NSCLC,most patient were diagnosed to advanced stage. Maintenance treatment is the continuation of treatment after first-line treatment and before the disease progresses. We consider to add apatinib,a tyrosine kinase inhibitor of VEGF,to the therapy of these patients. We designed the study to explore the possibility of apatinib for maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed of lung adenocarcinoma, EGFR wild-type or known drug-resistant mutation, stage IV or irradiative stage IIIB.
2. Age ≥ 18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1;
4. Patients had previously received at least 4 cycles of first-line, double chemotherapy and had no disease progression at baseline screening compared with baseline imaging prior to first-line chemotherapy；
5. Adequate hepatic, renal, heart, and hematologic functions: ANC ≥ 1.5×109/L, PLT ≥ 100×109/L, HB ≥ 90 g/L, TBIL ≤ 1.5×ULN, ALT or AST ≤ 2.5×ULN (or ≤ 5×ULN in patients with liver metastases), Serum Cr ≤ 1×ULN, Cr clearance ≥ 45 mL/min;

Exclusion Criteria:

1. Active brain metastases, meningococcal meningitis, patients with spinal cord compression, or imaging at CT or MRI examination revealed brain or pia mater disease（Patients who have completed treatment and whose symptoms are stable in the first 21 days of randomization may be enrolled in the study but may be diagnosed as having no intracerebral hemorrhage by MRI, CT or venography）；
2. Imaging (CT or MRI) showed that the tumor lesions were ≤ 5 mm from the major vessels or there was a central tumor invading local macrovascular；
3. Imaging (CT or MRI) showed significant cavitary or necrotic lung tumors, uncontrollable hypertension (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg, despite optimal medical therapy), grade II The above myocardial ischemia or myocardial infarction, poor control of arrhythmia (including QTc interval male ≥ 450 ms, female ≥ 470 ms); NYHA standards, Ⅲ ~ Ⅳ grade cardiac insufficiency, or cardiac ultrasound examination prompted left ventricular ejection Score (LVEF) <50%；
4. Coagulation dysfunction (INR> 1.5, PT> ULN +4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment；Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or the like；
5. Patients who had obvious hemoptysis within 2 months before screening, or experienced daily hemoptysis with a volume more than half a tea spoon (2.5ml) or above；
6. Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc.
7. Patients who manifested arterial/venous thrombus events, e.g. cerebrovascular accident (Including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening（Such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism and so on）；
8. Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g；
9. Confirmed ALK gene fusion；
10. Anti-angiogenic drugs were used during first-line chemotherapy。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause
Objective Response Rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Ma, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China